CLINICAL TRIAL: NCT06089629
Title: Frenuloplasty for Speech and Myofunctional Outcomes: a Randomized, Controlled Study
Brief Title: Frenuloplasty for Speech and Myofunctional Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Oregon Clinic (Other)
Responsible Party: Principal Investigator, Bobak Ghaheri, MD, Otolaryngologist, The Oregon Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Speech2023
Record Dates: First submitted 2023-10-08; First posted 2023-10-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Ankyloglossia; Speech Delay; Dentofacial Abnormalities
Keywords: ankyloglossia; speech delay; myofunctional therapy; dentofacial abnormalities
MeSH Terms: conditions — Ankyloglossia; Language Development Disorders; Dentofacial Deformities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Nonsurgical intervention with speech and myofunctional therapy
- Intervention group (Experimental): Surgical intervention with frenuloplasty followed by speech and myofunctional therapy
  Interventions: Procedure: Lingual frenuloplasty

INTERVENTIONS:
Procedure: Lingual frenuloplasty — Surgical release of ankyloglossia with suture reorientation of the wound to improve lingual mobility, done under local or general anesthesia
  Arms: Intervention group

SUMMARY:
Children with ankyloglossia (tongue tie) can have abnormal tongue function, putting them at a disadvantage when it comes to speech and articulation. Furthermore, abnormal tongue posture within the oral cavity increases the likelihood of myofunctional disorders.

DETAILED DESCRIPTION:
The current body of literature surrounding ankyloglossia and speed delay is mixed. The literature base is riddled with retrospective reviews, poor descriptions of surgical intervention, and the lack of standardized grading schemes with respect to articulation. Furthermore, the candidacy for intervention in these instances only involves children with anterior tongue tie. There is a complete lack of investigation surrounding the impact of posterior tongue tie on articulation.

The other area that has inadequately been studied is the impact ankyloglossia has on myofunctional outcomes. There are data now that demonstrate how ankyloglossia is correlated with a vaulted palate and has long term orthodontic consequences. This study aims to demonstrate how release of posterior tongue tie improves lingual strength and posture.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 5-12 with posterior tongue tie who are undergoing treatment just for ankyloglossia
* Children must already be working with an SLP who has done a speech and myofunctional evaluation

Exclusion Criteria:

* Children undergoing other procedures at the same time as the frenuloplasty (tonsillectomy, adenoidectomy, etc)
* Significant medical comorbidities (cardiovascular, neurological, etc)
* Anterior tongue tie or lip tie
* Previous lingual surgery

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Speech/Articulation | Baseline (timepoint 0) and 2 months post-intervention (surgical group) or 2 months post-therapy alone (control group)
  Using the GFTA-3 test of articulation
Tongue mobility | Baseline (timepoint 0) and 2 months post-intervention (surgical group) or 2 months post-therapy alone (control group)
  Using the TRMR grading scale
Tongue strength | Baseline (timepoint 0) and 2 months post-intervention (surgical group) or 2 months post-therapy alone (control group)
  Using the IOPI instrument

IPD SHARING:
Plan to Share IPD: No